CLINICAL TRIAL: NCT06122246
Title: PRESSURE CHECK: Find Your Path to Better Health
Acronym: PRESSURE CHECK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2000036141; HM-2022C2-28354 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Blood Pressure
Keywords: hypertension; remote patient monitoring; community health worker; digital health
MeSH Terms: conditions — Hypertension | interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: Community Based Organizations (CBO) will be randomized in a cluster-randomized stepped-wedge design in which CBOs will be randomized to one of 5 sequences.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remote Blood Pressure (BP) Management Program (Active Comparator): Participants are enrolled in a remote BP management program (RBPM) inclusive of home BP monitoring and telehealth visits with a nurse or pharmacist.
  Interventions: Other: Remote Blood Pressure (BP) Management Program (RBPM)
- Remote Blood Pressure (BP) Management Program + Community Health Worker (CHW) (Experimental): Participants are enrolled in a remote BP management program (RBPM) inclusive of home BP monitoring and telehealth visits with a nurse or pharmacist plus a social model with a CHW.
  Interventions: Behavioral: Community Health Worker (CHW); Other: Remote Blood Pressure (BP) Management Program (RBPM)
- Usual Care (No Intervention): Participants receive education about hypertension and are referred to primary care for ongoing management.

INTERVENTIONS:
Behavioral: Community Health Worker (CHW) — Participants will receive the additional support of a Community Health Worker (CHW).
  Arms: Remote Blood Pressure (BP) Management Program + Community Health Worker (CHW)
Other: Remote Blood Pressure (BP) Management Program (RBPM) — Participants will receive a medical model of remote BP management (RBPM).
  Arms: Remote Blood Pressure (BP) Management Program; Remote Blood Pressure (BP) Management Program + Community Health Worker (CHW)

SUMMARY:
This study seeks to develop the evidence for a sustainable, community-partnered, multi-level health system strategy to improve blood pressure control. Two team-based approaches are being tested: 1) a medical model of remote BP management (RBPM) alone, and 2) RBPM plus a social model with a community health worker (CHW). These 2 strategies are being compared with a standard community screening program with referral to primary care.

DETAILED DESCRIPTION:
In this comparative effectiveness trial, we aim to answer the research question of whether a remote blood pressure management program (RBPM, inclusive of home blood pressure monitoring and telehealth visits with a nurse or pharmacist) alone or an RBPM program with community health worker (CHW) support is more effective than standard screening with education and referral to primary care in controlling blood pressure and addressing social determinants that lead to poor health outcomes.

This is a multisite study using a stepped wedge design. Health systems in 4 different cities are each partnered with 10 community based organizations (CBOs). CBOs are randomized into one of 4 sequences. Each sequence moves through the 3 study arms at different time points: Community Standard, RBPM alone, and RBPM+CHW.

At the CBOs, research health advocates screen for hypertension. Qualifying individuals who provide informed consent can enroll in the study and are assigned to the intervention that the CBO is in at that particular time. All participants receive a blood pressure cuff and a device that syncs their data with the research database. If enrolled in the RBPM arm, participants are scheduled for telehealth visits with the Pressure Check medical team to improve blood pressure control through lifestyle support and medication initiation/titration. If enrolled in the RBPM+CHW arm, participants additionally receive support from a CHW to help with medical visits and address social determinants of health. The primary outcome is blood pressure control at 6 months. Additional outcomes include implementation science to understand factors associated with adoption and outcomes, and 12 and 18 month blood pressure control.

In partnering with the community, health systems can extend their reach. CBO leaders support health messaging around hypertension and increase trust between the health system and their clients (patients). The two models, RBPM alone and RBPM+CHW, are based on the concept that disparities in hypertension control among Black, Latinx, and low-income populations exist because of inequities related to health system access and trust, individual-level socioeconomic and lifestyle factors, the physical/built environment, sociocultural factors, and discriminatory policies. Addressing these barriers may improve blood pressure control.

ELIGIBILITY:
Inclusion Criteria:

* Elevated BP, defined as an average resting BP of >=135/85 mmHg based on 3 consecutive blood pressure readings

Exclusion Criteria:

* People who are pregnant
* Those that have end stage renal disease on dialysis
* People receiving active chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2024-04-14 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Control | 6 months
  Participants will be assessed at 6 months for Blood Pressure (BP) control- defined as BP <130/80 mmHg. To assess BP control, blood pressure will be measured in-person at the CBO (or another location) at Baseline, 6, 12 and 18 months with the primary endpoint of assessment as BP control at 6 months.

SECONDARY OUTCOMES:
Difference in systolic BP between study groups, measured at CBO | 6 months, 12 months, 18 months
  Mean difference in BP measured at CBO at baseline and follow-up; take average of last 2 of 3 measurements
Difference in BP control by study group, measured at CBO | 6 months, 12 months, 18 months
  Proportion of participants with BP with:
  Ideal <120/80 mmHg Intermediate: <=135/85 mmHg Poor: >135/85mmHg
Change in Well-being | 6 months, 12 months, 18 months
  Well-being is assessed with the 12-item 100 Million Healthier Lives. Cantrill's Ladder: stratification into Thriving, Suffering, Struggling. Will assess mean differences of 0.5 as meaningfully different
Change in Lifestyle behaviors | 6 months, 12 months, 18 months
  Differences in self-reported measures using a survey.Each measure is categorized as "ideal"(2 points), "intermediate"(1 point) or "poor" (0 point).

CONTACTS AND LOCATIONS:
Overall Officials: Erica Spatz, MD, Principal Investigator — Yale University; Rafael Perez-Escamilla, MD, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Yale, New Haven, Connecticut
  - Massachusetts General Brigham Hospital, Boston, Massachusetts
  - Houston Methodist, Houston, Texas
  - Sentara Health, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
After investigators complete the main reports, data will be shared upon request. When sharing data with other collaborators and the broader scientific community, all identifiers will be removed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared upon request.
Access Criteria: Because of the sensitive nature of the data collected in this study, investigators will require all users to enter into a data agreement that stipulates that 1) data will be used for research purposes only and will not be used to identify individual participants, 2) data will remain at Yale and a Yale analyst will run the requested data at the expense of the requestor. Under certain circumstances, we will transfer data to outside investigators after a DUA is signed.

REFERENCES:
- See also: Pressure Check website — https://www.pressurecheck.org/